CLINICAL TRIAL: NCT04404296
Title: Efficiency and Clinical Outcomes of 25-gauge, Bevel-tip, 20000 Cuts-per-minute, Pars Plana Vitrectomy
Brief Title: Pars Plana Vitrectomy With 25-gauge 20000 Cpm, Bevel-tip Cutter
Acronym: HYPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peregrine Eye and Laser Institute (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Harvey Siy Uy, Medical Director, Peregrine Eye and Laser Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190101
Record Dates: First submitted 2020-04-20; First posted 2020-05-27 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Vitrectomy; Retinal Detachment; Vitreous Hemorrhage; Macular Holes; Epiretinal Membrane; Dislocated Intraocular Lens Into Vitreous; Retained Lens Fragments
Keywords: Small gauge vitrectomy probe; 20000 cut per minute; Microincisional vitrectomy system
MeSH Terms: conditions — Retinal Detachment; Vitreous Hemorrhage; Retinal Perforations; Epiretinal Membrane

STUDY DESIGN:
Intervention Model Description: Interventional case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 25-gauge 20000 PPV (Other): Eyes will undergo pars plana vitrectomy using 25-gauge, bevel-tip, 20000 cut per minute vitrectomy probe
  Interventions: Device: 25-gauge, bevel-tip, 20000 cut per minute pars plana vitrectomy

INTERVENTIONS:
Device: 25-gauge, bevel-tip, 20000 cut per minute pars plana vitrectomy — Pars plana vitrectomy using 25-gauge, bevel-tip, 20000 cut per minute vitrectomy probe

SUMMARY:
Report efficiency and clinical outcomes using 25-gauge, bevel-tip, 20000 cut per minute vitrectomy probe among eyes with various vitreo-retinal diseases

DETAILED DESCRIPTION:
We will evaluate the efficiency and clinical outcomes of pars plana vitrectomy using a 25-gauge, bevel-tip, 10 and 20000 cpm vitrectomy probe among eyes with 8 main surgical indications. Main outcome measures included efficiency measures, postoperative pain and complications.

ELIGIBILITY:
Inclusion Criteria:

* All eyes undergoing pars plana vitrectomy with surgically amenable vitreoretinal disease.

Exclusion Criteria:

* History of prior PPV, glaucoma, scleral thinning, and active or recent history of (<3 months) ocular or extra-ocular infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Operative time: Total | 6 months
  From insertion of first trocar to removal of last trocar, measured in seconds using stopwatch

SECONDARY OUTCOMES:
Pain scoring | 6 months
  Visual Analogue scale (0 to 4)
Adverse events | Up to 3 months after surgery
  Intra- and Postoperative complications
Number of times ancillary instruments placed in eye | 6 months
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Uy, MD, Principal Investigator — Peregrine Eye and Laser Institute
Locations (1):
- Peregrine Eye and Laser Instittute, Makati City, MM, Philippines

IPD SHARING:
Plan to Share IPD: No